CLINICAL TRIAL: NCT06830408
Title: Swiss Cancer Registry on Safety and Efficacy of 177Lu-ITG-PSMA-1 Radionuclide Therapy in Prostate Cancer Patients
Brief Title: Performance of 177Lu-PSMA-I&T for RLT in mCRPC - Prospective Multicenter Swiss Registry Study
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: EKNZ 2021-01271
Record Dates: First submitted 2025-01-30; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: mCRPC
Keywords: radioligand therapy; 177Lu-PSMA-I&T; registry-study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient wit progressive mCRPC
  Interventions: Drug: radionuclide therapy with 177Lu-PSMA-I&T

INTERVENTIONS:
Drug: radionuclide therapy with 177Lu-PSMA-I&T — Standard PSMA RLT with 7-8 GBq i.v. infusion of 177Lu-PSMA-I&T performed every 6-8 weeks for 4-6 cycles, or until progression or complete response.

SUMMARY:
The goal of this observational study (multicenter, national registry-based) is to evaluate the performance of 177Lu-ITG-PSMA-1 (177Lu-PSMA-I&T) as therapy in patients with metastatic castration resistent prostate cancer (mCRPC).

The main questions are whether the 177Lu-PSMA-I&T is safe and if it works well to treat patients with progressive mCRPC. The data and information in the study are collected under standard medical therapy and follow-up, so called real-world conditions.

Participants will:

* undergo regular radioligand therapy (RLT) with 177Lu-PSMA-I&T
* have clinical, laboratory and imaging follow-up according to the currently available recommendation for PSMA-RLT an in line with their medical needs.
* answer study related set of questionnaires

DETAILED DESCRIPTION:
Prospective, multicenter Swiss registry study evaluating the performance of 177Lu-ITG-PSMA-1 (177Lu-PSMA-I&T) as RLT in mCRPC.

Primary endpoint: Safety-

* frequency and severity of adverse events (measured according to CTCAE 5.0). Secondary endpoints: Efficacy
* biochemical response: best PSA response, PSA50 (>50% decrease from baseline PSA level) and PSA response at 12 weeks

  * imaging response: Objective response rate evaluated on follow-up morphological imaging CT/MRI and/or on molecular imaging PSMA PET/CT
  * quality of life: evaluated with standardized questionnaires

ELIGIBILITY:
Inclusion Criteria:

* hormone-refractory and PSMA PET/CT-positive prostate tumors
* progressed after or are ineligible for chemotherapy, next-generation antihormonal therapy or bone-directed radiation therapy -- male patients with an age above 18 years

Exclusion Criteria:

* patients who are not eligible for PSMA RLT, according to current, standard medical indications and guidelines
* patients who for medical or non-medical reasons are unable to give their consent
* patients withdrawing their consent for participation (NB: the already collected data in such cases will be anonymized and further used for applicable analyses)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with progressive mCRPC who are eligible for PSMA RLT
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2025-01-13 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of treatment related adverse event | performed at baseline (before starting the first therapy cycle), during (before each additional therapy cycle) and at 8-14 weeks after completion of all therapy cycles
  frequency and severity of treatment related adverse events evaluated on standard blood tests (CBC, liver and kidney function)-, according to CTCAE 5.0

SECONDARY OUTCOMES:
Efficacy - biochemical response | performed at baseline (before starting the first therapy cycle), during (before each additional therapy cycle) and at 8-14 weeks after completion of all therapy cycles
  -measured by changes from baseline PSA (ng/ml), according to the PCWG3
Efficacy - imaging response | PSMA PET/CT performed at baseline (before starting the first therapy cycle), PSMA SPECT/CT during therapy (24-48 hours after each cycle) and PSMA PET/CT (and/or CT/MRI) at 8-14 weeks after completion of all therapy cycles
  objective response rates from, evaluated on morphological imaging according to RECIST criteria and on molecular imaging according to the Consensus statements on PSMA PET/CT response assessment criteria
Quality of life - EORTC PR25 | performed at baseline, before each therapy cycle and at 8-14 weeks after completion of all therapy cycles
  evaluated with the standardized EORTC PR25 questionnaire
Quality of life - pain | performed at baseline, before each therapy cycle and at 8-14 weeks after completion of all therapy cycles
  evaluated with the standardized Brief Pain Inventory
Quality of life - Xerostomia | performed at baseline, before each therapy cycle and at 8-14 weeks after completion of all therapy cycles
  evaluated with the standardized Xerostomia questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Alin Chirindel, Principal Investigator — University Hospital, Basel, Switzerland
Locations (8):
- Switzerland (8):
  - University Hospital Basel, Basel, Canton of Basel-City
  - CHUV, Lausanne, Canton of Vaud
  - Kantonspital Aarau, Aarau
  - Inselspital, Bern
  - Luzerner Kantonsspital, Lucerne
  - St. Anna Hirslanden Klinik, Lucerne
  - Kantonsspital St. Gallen, Sankt Gallen
  - University Hospital Zurich, Zurich